CLINICAL TRIAL: NCT01666392
Title: The Impact of Omega-3 Fatty Acid Supplementation on Markers of Inflammation and Lean Body Mass in Older Adults
Brief Title: Omega-3 Fatty Acid Supplementation in Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Nordic Naturals (Industry)
Responsible Party: Principal Investigator, Zsolt Murlasits, Assistant Professor, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: #2232; #2232 (Other: The University of memphis)
Record Dates: First submitted 2012-08-10; First posted 2012-08-16 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-08

CONDITIONS: Inflammation
Keywords: Omega-3 fatty acid; Fish oil; Muscle mass; Muscle strength; Older adults; Circulating inflammatory cytokines; Skeletal muscle mass; Upper body strength; Lower body strength
MeSH Terms: conditions — Inflammation | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Omega-3 fatty acid) (Experimental): 2 capsules/day of ProOmega providing 650mg EPA and 450mg DHA
  Interventions: Dietary Supplement: Omega-3 fatty acid
- Soybean oil (Placebo Comparator): 2 capsules/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — Omega-3 fatty acid, Eicosapentaenoic acid+docosahexaenoic acid in capsule form
  Other Names: ProOmega (Nordic Naturals)
  Arms: Fish oil (Omega-3 fatty acid)
Dietary Supplement: Placebo — Placebo
  Arms: Soybean oil

SUMMARY:
The purpose of this study to determine whether Fish oil (Omega-3 Fatty Acid) supplementation has an impact on inflammation and lean body mass in older adults. The investigators expect that Fish oil supplementation will reduce inflammation and prevent the loss of lean mass compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or over

Exclusion Criteria:

* Fish, seafood allergies, nut allergies, soy allergies
* Habitual (>1/week) fish or seafood consumption
* Current Omega-3 supplement use
* Gastrointestinal problems
* Current anti-inflammatory medication use
* Current anticoagulant medication use

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
C-Reactive protein | At baseline testing and at 3 month endpoint
  Inflammatory marker
IL6 | At baseline and at 3 month endpoint
  Inflammatory cytokine
TNFα | At baseline and at 3 month endpoint
  Inflammatory cytokine

SECONDARY OUTCOMES:
Skeletal muscle mass/body composition | At baseline testing and at 3 month endpoint
  The amount of skeletal muscle mass and fat mass and their ration will be determined.
Lower body muscular strength | At baseline and at 3 month endpoint
  Measurement of maximum strength in the leg press exercise
Upper body muscular strength | At baseline and at 3 month endpoint
  Measurement of maximum strength in the chest press exercise

OTHER OUTCOMES:
EPA and DHA | At baseline and at 3 month endpoint
  To determine the effectiveness of fish oil supplementation, we measure EPA and DHA Omega-3 fatty acid levels

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Murlasits, Ph.D., Principal Investigator — The University of Memphis
Locations (1):
- Department of Health and Sport Sciences, The University of Memphis, Memphis, Tennessee, United States